CLINICAL TRIAL: NCT03585777
Title: Serum Klotho Level in Patients on Oral Antidiabetic Treatment
Brief Title: Compare Serum Klotho Levels in Patients on Oral Antidiabetic Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelkawi Hammad, Lecturer of internal medicine,faculty of medicine,Fayoum university, Fayoum University
Other Study IDs: VCG 3
Record Dates: First submitted 2018-02-09; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Compare Serum Level of Klotho in Patients on Oral Antidiabetic Treatment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Compare serum levels of klotho in patients taking glimepiride in comparison to patients taking metformin
- Group 2: Compare serum levels of klotho in patients taking glimepiride in comparison to patients taking linagliptin
- Group 3: Compare serum levels of klotho in patients taking glimepiride in comparison to patients taking impaglifluzin

SUMMARY:
Klotho is a protein found in serum, kidney,heart,brain and in other tissues,it has many functions,it is viewed as the anti aging hormone. Aging kidneys are characterized by progressive scarring and measurable declines in renal function

DETAILED DESCRIPTION:
Objectives To study serum klotho level among diabetic patients attending diabetes and endocrine clinic in Fayoum university on oral antidiabetic treatment

Study Design:

This study will be an observational prospective cohort study. The study duration will be 2 months.

Study Methods:

* Population of Study
* Group 1 :compare serum klotho levels in patients taking glimeperirde versus levels in patients taking metformin
* Group 2 : compare serum klotho levels in patients taking glimeperirde versus levels in patients taking linagliptin
* Group 3 : compare serum klotho levels in patients taking glimeperirde versus levels in patients taking impaglifluzin
* Inclusion Criteria :
* Group 1 :Diabetics candidate for oral treatment
* Group 2 :Diabetics candidate for oral treatment
* Group 3 :Diabetics candidate for oral treatment
* Exclusion Criteria :

Diabetics candidate for insulin treatment

There will be three arms to this study; the first arm will enroll patients on glimepiride and patients on metformin to compare serum klotho levels. The second arm will enroll patients on glimepiride and patients on linagliptin to compare serum klotho levels. The third arm will enroll patients on glimepiride and patients on impaglifluzin to compare serum klotho levels Each arm will enroll 40 patients, 20 patients on glimiperide treatment,20 patient will on the other drug,patients will be selected from Fayoum university diabetes and endocrine clinic

Data collection:

Patients will be subjected to; full clinical examination,waist hip ratio assessment,BMI assessment fasting blood glucose,2PP blood glucose,HbA1C, urea, creatinine, uric acid total calcium,albumin, phospherus, estimated GFR, ACR, total cholesterol, triglycerides, serum klotho, FGF 23 levels assessment , also fracrtional excretion of phospherus will be assessed. Control of blood glucose will be done along the period of the study. At the end of the 2 months,reassessment of the above mentioned parameters will be done.

ELIGIBILITY:
Inclusion Criteria:

* Diabetics candidate for oral treatment

Exclusion Criteria:

* Diabetics candidate for insulin treatment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetics on oral treatment
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-10-11 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Beneficial effect manifested by a statistical significant decrease in klotho levels | 2 months
  An anticipated statistical significant decrease in klotho level

SECONDARY OUTCOMES:
No beneficial effect manifested by by a non significant decrease in klotho level or a rise in the level | 2 months
  Non statistical significant decrease in klotho level, or a significant rise in it

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum university Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided